CLINICAL TRIAL: NCT07134725
Title: Phase 1/2, Double-blind, Randomized, Active-controlled First-in-human Clinical Trial to Evaluate the Safety and Immunogenicity of the Chimeric SpiN-Tec MCTI UFMG Vaccine for Covid19
Brief Title: Safety and Immunogenicity of a Chimeric Recombinant Covid19 Vaccine SpiN-Tec MCTI UFMG
Acronym: SpiN-Tec-001
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Federal University of Minas Gerais (Other)
Collaborators: Oswaldo Cruz Foundation (Other); The Ministry of Science, Technology and Innovation, Brazil (Unknown); Prefeitura de Belo Horizonte (PBH) (Unknown)
Responsible Party: Principal Investigator, Helton da Costa Santiago, Study Director, Federal University of Minas Gerais
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: SpiN-Tec-001; U1111-1300-1526 (Other: WHO International Clinical Trials Registry Plataforms); 5.536.100 (Other: Ethics Committee of the Federal University of Minas Gerais); 5.569.964 (Other: Brazilian Ethics Committee (CONEP)); 59871822.1.1001.5149 (Other: Plataforma Brasil)
Record Dates: First submitted 2025-08-19; First posted 2025-08-21 (Actual); Last update posted 2025-09-15 (Actual); Status verified 2025-09

CONDITIONS: COVID - 19
Keywords: vaccine; infectious; viral disease; SARS-Cov-2; Coronavirus Infections; Coronavirus Disease 2019; Respiratory Tract Infections
MeSH Terms: conditions — COVID-19; Communicable Diseases; Virus Diseases; Coronavirus Infections; Respiratory Tract Infections

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (9):
- Phase 1 - arm 1: 20 ug SpiN-Tec (Experimental): 9 participants aged 18 to 54 years receiving 1 dose of the SpiN-Tec MCTI UFMG vaccine with 20 micrograms.
  Interventions: Biological: SpiN-Tec MCTI UFMG
- Phase 1 - arm 2: 60 ug SpiN-Tec (Experimental): 9 participants aged 18 to 54 years receive 1 dose of the SpiN-Tec MCTI UFMG vaccine with 60 micrograms.
  Interventions: Biological: SpiN-Tec MCTI UFMG
- Phase 1 (Active Comparator): 6 participants (3 participants in the age group of 18 to 54 years and 3 participants in the age group of 55 to 85 years ) will receive 1 dose of the active comparator
  Interventions: Other: Active Comparator: Covishield® vaccine
- Phase 2: 60 ug SpiN-Tec (Experimental): reinforcement with 60 ug of SpiN-Tec MCTI UFMG, 180 individuals, 30% of whom are between 55 and 85 years old.
  Interventions: Biological: SpiN-Tec MCTI UFMG; Other: Active Comparator: Comirnaty® vaccine
- Phase 2 (Active Comparator): reinforcement with active comparator, 180 individuals, 30% from the age group between 55 and 85 years old.
  Interventions: Other: Active Comparator: Comirnaty® vaccine
- Phase 1 - arm 3: 100 ug SpiN-Tec (Experimental): 9 participants aged 18 to 54 years receive 1 dose of the SpiN-Tec MCTI UFMG vaccine with 100 micrograms.
  Interventions: Biological: SpiN-Tec MCTI UFMG
- Phase 1 - arm 1b: 20 ug SpiN-Tec (Experimental): 9 participants aged 55 to 85 years receiving 1 dose of the SpiN-Tec MCTI UFMG vaccine with 20 micrograms.
  Interventions: Biological: SpiN-Tec MCTI UFMG
- Phase 1 - arm 2b: 60 ug SpiN-Tec (Experimental): 9 participants aged 55 to 85 years receive 1 dose of the SpiN-Tec MCTI UFMG vaccine with 60 micrograms.
  Interventions: Biological: SpiN-Tec MCTI UFMG
- Phase 1 - arm 3b: 100 ug SpiN-Tec (Experimental): 9 participants aged 55 to 85 years receive 1 dose of the SpiN-Tec MCTI UFMG vaccine with 100 micrograms.
  Interventions: Biological: SpiN-Tec MCTI UFMG

INTERVENTIONS:
Biological: SpiN-Tec MCTI UFMG — Chimeric recombinant protein (SpiN) adjuvanted with CTVad1
  Arms: Phase 1 - arm 1: 20 ug SpiN-Tec; Phase 1 - arm 1b: 20 ug SpiN-Tec; Phase 1 - arm 2: 60 ug SpiN-Tec; Phase 1 - arm 2b: 60 ug SpiN-Tec; Phase 1 - arm 3: 100 ug SpiN-Tec; Phase 1 - arm 3b: 100 ug SpiN-Tec; Phase 2: 60 ug SpiN-Tec
Other: Active Comparator: Covishield® vaccine — active comparator using vaccine approved by ANVISA (Brazilian Health Regulatory Agency)
  Arms: Phase 1
Other: Active Comparator: Comirnaty® vaccine — active comparator using vaccine approved by ANVISA (Brazilian Health Regulatory Agency)
  Arms: Phase 2; Phase 2: 60 ug SpiN-Tec

SUMMARY:
SpiN-Tec MCTI UFMG will be used as a vaccine booster against COVID-19 and will be evaluated using the active comparator, a vaccine approved by ANVISA (Brazilian Health Regulatory Agency). The study will consist of two parts: Part A) a Phase 1 dose-escalation clinical trial to assess safety and reactogenicity; followed by Part B) a Phase 2 clinical trial to assess the safety and immunogenicity of SpiN-Tec. The study will include healthy participants of both sexes, aged 18 to 85, who have already received the full COVID-19 vaccination schedule with CoronaVac® (Butantan) or Covishield® (AstraZeneca) and who have received one or two booster doses of Covishield® or Comirnaty® (Pfizer's RNA-based vaccine) at least 6 months ago. Participants may or may not have had natural SARS-CoV-2 infection.

DETAILED DESCRIPTION:
SpiN-Tec-001 is a multicenter, double-blind, randomized, controlled with active comparator (Covishield®), escalating dose study to verify the safety and immunogenicity of the investigational product, SpiN-Tec MCTI UFMG. SpiN-Tec MCTI UFMG is a heterologous vaccine booster and will be evaluated using the active comparator, Covishield® (AstraZeneca), as a reference, which will be the homologous or heterologous booster to the primary vaccination. The study will consist of two parts: Part A) a phase 1 dose-escalation clinical trial to verify the safety and reactogenicity of the investigational product, followed by Part B) a phase 2 clinical trial to study the safety and immunogenicity of SpiN-Tec. The study intends to evaluate a booster dose with the SpiN-Tec MCTI UFMG vaccine in healthy participants of both sexes who have already received the complete vaccination schedule for COVID-19 with the CoronaVac® (Butantan) or Covishield® ( AstraZeneca) and who have received one or two booster doses of Covishield® or Comirnaty® (Pfizer's RNA-based vaccine) for at least 6 months. Participants may or may not have had a natural infection with SARS-CoV-2. The participants' last antigenic stimulation (boost or infection) must have occurred at least 6 months before randomization in the study. Part A (Phase 1): double-blind, randomized (within the same arm) clinical trial in an escalating dose and controlled with an active comparator to verify the safety of SpiN-Tec MCTI UFMG. For this part, participants who have completed the vaccination schedule with CoronaVac® and have received a single booster dose with Comirnaty® (Pfizer) between 9 and 15 months of inclusion and who have no history of COVID-19. The study includes 24 participants in each of the 3 arms, based on the doses of SpiN-Tec MCTI UFMG, and each arm consists of two age groups. Furthermore, this is a sentinel group within each arm: Arm 1 - 20 µg of SpiN-Tec MCTI UFMG (N=18) or active comparator (N=6): 18 participants (9 participants aged 18 to 54 years and 9 participants in the age group of 55 to 85 years) receiving 1 dose of the SpiN-Tec MCTI UFMG vaccine with 20 micrograms and 6 participants (3 participants in the age group of 18 to 54 years and 3 participants in the age group of 55 to 85 years ) will receive 1 dose of the active comparator. The sentinel group is the first three individuals recruited from the youngest age group. Two of these individuals received SpiN-Tec MCTI UFMG, and the other individual, the active comparator, was randomized blindly and observed for at least 7 days before continuing vaccination in the corresponding age group. Arm 2 - 60 µg of SpiN-Tec MCTI UFMG (N=18) or active comparator (N=6): 18 participants (9 participants aged 18 to 54 years and 9 participants aged 55 to 85 years) receive 1 dose of the SpiN-Tec MCTI UFMG vaccine with 60 micrograms and 6 participants (3 participants aged 18 to 54 years and 3 participants in the age group 55 to 85 years) will receive 1 dose of the active comparator. The sentinel group is the first three individuals recruited from the youngest age group. Two of these individuals receive SpiN-Tec MCTI UFMG, and the other individual, the active comparator, is blindly randomized and observed for at least 7 days before continuing vaccination in the corresponding age group. Arm 3 - 100 µg SpiN-Tec MCTI UFMG (N=18) or active comparator (N=6): 18 participants (9 participants aged 18 to 54 years and 9 participants aged 55 to 85 years) receive 1 dose of the SpiN-Tec MCTI UFMG vaccine with 100 micrograms and 6 participants (3 participants aged 18 to 54 years and 3 participants aged 55 to 85 years) will receive 1 dose of the active comparator. The sentinel group is the first three individuals recruited from the youngest age group. Two of these individuals receive SpiN-Tec MCTI UFMG, and the other individual, the active comparator, is blindly randomized and observed for at least 7 days before continuing vaccination in the corresponding age group. All participants in the sentinel cohorts in Part A are under observation at the Research Center for at least 60 minutes after vaccine administration. The remaining participants are under observation for at least 30 minutes. All participants in Part A are monitored for 360 days with regular clinical assessments through Telephone contact on days 1, 3, 10, and 21 and then monthly until the end of the study, except when there is an in-person visit. The sentinel cohort has additional contact on day 5. In-person return on days 7, 14, 28, 90, 180, 270 and 360 after vaccination. Participants are recruited and allocated sequentially to arms 1, 2, and 3 of the study, respectively receiving doses of 20 ug, 60 ug, and 100 ug of the investigational product, and, in each age group of each arm, 9 participants receive the SpiN-Tec MCTI UFMG vaccine and 3 active comparator, totaling 12 participants for the younger age group (18-54 years) and 12 participants for the older age group (55-85 years). Of these, 18 participants received reinforcement with SpiN-Tec MCTI UFMG, and 6 received reinforcement with the active comparator. The first group recruited volunteers aged 18 and 54 to administer the lowest dose (20 µg) of SpiN-Tec MCTI UFMG. The first three randomized subjects in this age group are the sentinel group and observed for at least 7 days before continuing vaccination in that arm.

Adverse events (AEs) of the sentinel cohort are evaluated by the protocol and safety review team (TRPS) within 7 days of vaccination, and if no study suspension criteria are met, vaccination for the remainder of the arm is proceeded. After the first 14 days of follow-up for all individuals in this age group, a new blinded safety analysis will be carried out by TRPS for the dose and age group escalation decision. If no criteria for suspension of the study are found, the TRPS must recommend continuing the study. If any criterion for stopping the study is observed, or if a member of the TRPS deems it necessary, a meeting with an independent safety monitoring committee (CIMS) must be requested. If consulted, CIMS will receive the safety data and must recommend continuing the study as planned, suggesting changes to the protocol, or recommending stopping the study. This procedure must be repeated for each dose escalation or age group. If the TRPS recommendation is to continue the study, volunteers from the same arm aged between 55 and 85 years will be randomized. Likewise, individuals between 18 and 54 in Arm 2 (60 ug of SpiN-Tec MCTI UFMG) will be vaccinated, with the first three individuals in Arm 2 making up the sentinel cohort and will be observed for 7 days before continuing randomization of that same arm. After completion of the first 14 days of follow-up in the youngest age group of Arm 2, a safety analysis by TRPS will be performed to decide on dose escalation (Arm 3) and age group 55-85 years (Arm 2). Likewise, the first three subjects in Arm 3 will be from the sentinel cohort and observed for 7 days before continuing vaccinations in that arm. Before lane escalation for Arm 3, a TRPS safety analysis must be carried out, as occurred in the other arms. At the end of the V28 visit of the last randomized participant in Part A, a blinded interim analysis of safety data and preliminary immunogenicity data (neutralizing antibodies against the ancestral strain and relevant VoCs at the time of the study, binding antibodies and IFNg production) should be performed and carried out before the study continued. CIMS will receive safety and preliminary immunogenicity data for analysis.

The Sponsor will suggest a dose for Part 2 of the study based on safety data and preliminary immunogenicity data that the study Scientific Committee and CIMS must previously approve. The dose with the best preliminary immunogenicity performance associated with the lowest intensities and frequencies of AEs will be chosen. Part B: after the interim analysis of the results obtained in Part A and approval by ethical regulatory bodies, the chosen dose of SpiN-Tec MCTI UFMG will be used as a vaccine booster for participants in the experimental arm of Part B of the study. The vaccination booster is very advanced in Brazil, reaching more than 80% of the population vaccinated so far (September 2022), and could be at even higher levels when the study begins. Therefore, recruitment will seek to include individuals who have received a booster (either one or two doses). Thus, in this study phase, an additional 180 participants who will receive the SpiN-Tec MCTI UFMG vaccine will be recruited, and another 180 participants will receive the active comparator. At least 30% of Part B participants must be between 55 and 85. Therefore, the study arms in Part B will be: Arm 1: reinforcement with SpiN-Tec MCTI UFMG, 180 individuals, 30% of whom are between 55 and 85 years old. Arm 2: reinforcement with Covishield®, 180 individuals, 30% from the age group between 55 and 85 years old. All participants in Part B will be under observation at the Research Center for at least 30 minutes after vaccine administration and will be monitored for 360 days with regular clinical assessments through Telephone contact on days 1, 3, 10, 21, and then monthly until the end of the study, except in the months when there will be an in-person visit. In-person return on days 7, 14, 28, 90, 180, 270 and 360 after vaccination. Therefore, the study will recruit a total of 432 participants, with 72 participants in Part A and 360 participants in Part B. After all participants in Part B complete 70 days of follow-up after the vaccine, after contact C70, there will be a break in the blinding and analysis of safety and immunogenicity data to verify the primary outcome of Part B. From that point on, the study is no longer double-masked, and participants continue to be monitored for safety purposes.

ELIGIBILITY:
Inclusion Criteria:

Part A: Healthy individuals aged 18 to 54 with completed primary vaccination schedule for COVID-19 with CoronaVac®. Have received a booster dose with Comirnaty® between 9 and 15 months before inclusion in the study.

Part A2: Healthy individuals aged 55 to 85 with a completed vaccination schedule for COVID-19 with CoronaVac® or Covishield® for at least six months from inclusion in the study. Have received at least one booster dose with Comirnaty® or Covishield® at least six months ago.

Part B: Healthy individuals aged 18 to 85 who completed the vaccination schedule for COVID-19 with CoronaVac® or Covishield® for at least six months from inclusion in the study. Have received at least one booster dose with Comirnaty® or Covishield® at least six months ago.

All Parties:

* Consent to the study and its procedures, documented by signing the Free and Informed Consent Form (TCLE).
* Present good general health as determined by medical examination.
* Agree not to donate blood while participating in the study.
* Women of childbearing potential must agree to use acceptable contraception* for at least 30 days before initiation of vaccination and at least 90 days following the use of the investigational product or active comparator.

  * Acceptable contraceptive methods: Barrier methods, including condoms or cervical caps. Surgically sterile partner/participant (including those undergoing vasectomy, hysterectomy, bilateral oophorectomy, and or tubal ligation) who is the only partner. Intrauterine device (with or without hormones) implanted. Birth control medications (oral, topical, injectable, or implantable). True sexual abstinence is in line with the patient's preferred and usual lifestyle. Note: periodic abstinence, such as calendar, ovulation, symptothermal, post-ovulation, or coitus interruptus methods, will not be considered a valid method.

Exclusion Criteria:

Part A:

* No previous history or acute infection with SARS-CoV-2. Previous records will be considered self-declaration by the participant.
* Vaccination booster for COVID-19 less than nine months ago and more than 15 months after inclusion in the study.
* The presence of comorbidities or any condition that, in the study investigator's assessment, could put the participant at risk or create a confounding factor in the study, including clinically stable chronic diseases.

Part A2:

* Acute SARS-CoV-2 infection or less than six months from the date of inclusion in the study.
* Vaccination booster for COVID-19 less than six months ago.
* The presence of comorbidities or any condition that, in the study investigator's assessment, could put the participant at risk or create a confounding factor in the study, including clinically stable chronic diseases.

Part B:

* Acute or SARS-CoV-2 infection or less than six months from the date of inclusion.
* Vaccination booster for COVID-19 less than six months ago.
* Any condition that, in the assessment of the study investigator, could put the participant at risk or create a confounding factor in the study. Diseases such as diabetes, hypertension, and clinically stable neuralgia may not constitute an exclusion criterion as determined by the medical investigator.

All Parties:

* Have received primary vaccination with Janssen or Comirnaty® vaccine.
* Have received a booster vaccine with the Janssen or CoronaVac® vaccine.
* History of SAE after administration of a COVID-19 vaccine.
* History of thrombophilia.
* Being on anticoagulant therapy or having a bleeding disorder that contraindicates intramuscular injection.
* Positive serology for HIV, HBV (HBsAg) or HCV.
* Laboratory abnormality in blood count, biochemistry, or urine tests. Exception will be defined by the clinical investigator when evaluated together with the participant's medical history.
* Women who are pregnant, breastfeeding, or intend to become pregnant/breastfeed within three months of inclusion in the study.
* Evidence of clinically active disease such as, but not limited to: neurological, renal, cardiovascular, endocrine, pulmonary, hepatic, hematological, immunological (including autoimmunities and immunodeficiencies), neoplastic or infectious disease.
* Psychiatric illness or cognitive impairment that, in the investigator's judgment, may affect the participant's ability to engage in the clinical trial following the established agenda.
* Alcohol abuse or use of illicit drugs in the last 12 months before recruitment has caused any family, medical, or professional problems.
* History of severe allergic reaction or anaphylaxis to any component of the vaccine.
* History of asplenia.
* Have participated in any other experimental clinical trial in the 12 months before inclusion or intend to participate in any experimental clinical trial in the 12 months following participation.
* Plans to participate in other clinical studies concurrently with this one. Use of some immunosuppressive therapy three months before recruitment or planning its use within three months after vaccination, including use of corticosteroids or other immunosuppressive medication (note: the immunosuppressive dose of corticosteroids is equivalent to 20 mg/day of prednisone per more than a week (topical or nasal corticosteroids are not considered immunosuppressive).
* Use of blood products (blood or immunoglobulins) within three months before inclusion or indication of their use during the study.
* Suspected active infection or confirmed fever (axillary temperature ≥ 38.0 oC) within 72 hours before inclusion. Recruitment should be delayed until the participant remains fever-free for 72 hours.
* Have received any live attenuated or inactivated vaccine within 28 days or 14 days, respectively, before use of the investigational product or active comparator or planning immunization within 28 days of study inclusion.
* History of use of medication authorized by ANVISA intended to prevent or treat COVID-19 less than six months before the study's inclusion date.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 432 (Actual)
Dates: Start 2022-11-23 (Actual); Primary Completion 2023-05-22 (Actual); Study Completion 2025-05-07 (Actual)

PRIMARY OUTCOMES:
Parts A, A2 e B: safety and reactogenicity for EAG and EAIE | In the first 28 days to EAG and EAIE for the entire duration of the study after immunization
  A, A2 e B: the investigators expect to evaluate the safety and reactogenicity for spontaneous adverse events in the first 28 days to EAG and EAIE for the entire duration of the study after intramuscular administration of SpiN-Tec MCTI UFMG as a booster in vaccination for COVID-19 through the evaluation of the frequencies (absolute and relative) and summary measurements (such as median and interquartile range), to describe qualitative variables (requested and unsolicited clinical AEs) and quantitative (laboratory AEs, size of erythema and edema, degree of AEs ), respectively, used to verify whether the outcome occurred
Part A: define a safe and immunogenic dose of SpiN-Tec MCTI UFMG to be used in Part B | At the end of visit V28 of the last randomized participant in Part A
  A: the investigators expect to define a safe and immunogenic dose of SpiN-Tec MCTI UFMG to be used in Part B of the study through the results of frequencies (absolute and relative) and summary measures (such as median and interquartile range), with the aim of to describe qualitative variables (solicited and unsolicited clinical AEs) and quantitative variables (laboratory AEs, size of erythema and edema, degree of AEs), respectively; post-baseline levels of neutralizing antibodies, binding antibodies and IFNg production will be calculated for each dose; and the increment of the parameters of each arm will be compared with the other dose-arms of the study.
Parte B: prove the non-inferiority of SpiN-Tec MCTI UFMG in inducing neutralizing antibodies | On day 28 after the booster of the SpiN-Tec MCTI UFMG vaccine
  B: the investigators expect to prove the non-inferiority of SpiN-Tec MCTI UFMG in inducing neutralizing antibodies will be verified by the geometric mean ratio of the increase in neutralizing antibody titers against the ancestral strain and against relevant VOCs at the time of the study on day 28 after the booster of the SpiN-Tec MCTI UFMG vaccine compared to the active comparator by evaluating the geometric mean increase in neutralizing antibody titers on a logarithmic scale induced by SpiN-Tec MCTI UFMG will be compared to the geometric mean increase in neutralizing antibody titers (baseline change) on a logarithmic scale generated by Covishield®. A 15% non-inferiority margin will be considered a parameter for neutralizing antibody levels.

SECONDARY OUTCOMES:
Parts A and A2: identify an increase in the levels of neutralizing antibodies | On days 14, 28, 90, 180, 270, and 360 after the booster
  A and A2: the investigators expect to identify an increase in the levels of neutralizing antibodies induced by SpiN-Tec MCTI UFMG measured by the geometric mean of neutralizing antibody titers on days 14, 28, 90, 180, 270, and 360 after the booster with the SpiN- Tec MCTI UFMG against time 0, measured by post-baseline levels of neutralizing antibodies to the ancestral strain and each relevant VoCs.
Parts A and A2: observe an increase in the average levels of anti-S, anti-RBD, and anti-N IgG antibodies | On days 14, 28, 90, 180, 270, and 360 after the booster
  A and A2: the investigators expect to observe an increase in the average levels of anti-S, anti-RBD, and anti-N IgG antibodies, measured by the geometric mean (in U/mL), on days 14, 28, 90, 180, 270, and 360 after the booster with the SpiN-Tec MCTI UFMG vaccine compared to time 0 measured by post-baseline antibody levels will be calculated for each participant and each evaluated antigen.
Parts A and A2: observe an increase in the IFNg levels in response to S and N antigens | On days 14, 28, 90, 180, 270, and 360 after the booster
  A and A2: the investigators expect to observe an increase in the geometric mean of IFNg levels (in pg/mL) produced by PBMCs in response to S and N antigens on days 14, 28, 90, 180, 270, and 360 after the SpiN-Tec vaccine booster MCTI UFMG compared to time 0 measured by post-baseline levels of antibodies calculated for each participant and for each evaluated antigen.
Part B: show an increase in the neutralizing antibody titers, in the levels of anti-S, anti-RBD, anti-N IgG, and anti-VoCs IgG antibodies, and an increase in the in IFNg levels. | On days 14, 28, 90, 180, 270 and 360 after the booster
  B: The SpiN-Tec MCTI UFMG vaccine is expected to show a Geometric Mean increase in neutralizing antibody titers, an increase in the levels of anti-S, anti-RBD, and anti-N IgG antibodies, and anti-VoCs IgG antibodies, and an increase in the geometric mean of the rise in IFNg levels produced by PBMCs stimulated with S and N antigens on days 14, 28, 90, 180, 270 and 360 after boosting with the SpiN-Tec MCTI UFMG vaccine compared to time 0 measured by ELISA assay.

CONTACTS AND LOCATIONS:
Overall Officials: Ricardo T Gazzinelli, DVM, PhD, Study Chair — Vaccine Technology Center (CT Vacinas)
Locations (1):
- Faculdade de Medicina da UFMG - Unidade de Pesquisa Clínica em Vacinas (UPqVac), Belo Horizonte, Minas Gerais, Brazil

IPD SHARING:
Plan to Share IPD: Undecided
The investigators are currently assessing the feasibility of sharing IPD, considering ethical, legal, and institutional requirements. A final decision has not yet been made.

REFERENCES:
- [Background] Hojo-Souza NS, de Castro JT, Rivelli GG, Azevedo PO, Oliveira ER, Faustino LP, Salazar N, Bagno FF, Carvalho AF, Rattis B, Lourenco KL, Gomes IP, Assis BRD, Piccin M, Fonseca FG, Durigon E, Silva JS, de Souza RP, Goulart GAC, Santiago H, Fernandes APS, Teixeira SR, Gazzinelli RT. SpiN-Tec: A T cell-based recombinant vaccine that is safe, immunogenic, and shows high efficacy in experimental models challenged with SARS-CoV-2 variants of concern. Vaccine. 2024 Dec 2;42(26):126394. doi: 10.1016/j.vaccine.2024.126394. Epub 2024 Oct 4. PMID 39368129